CLINICAL TRIAL: NCT05915988
Title: Wireless Ultra Long-Term EEG Recordings in Epilepsy - A Prospective Long-term Clinical Evaluation Using the UNEEG EpiSight Solution
Brief Title: U011 - Wireless Ultra Long-Term EEG Recordings in Epilepsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNEEG Medical A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UNEEG-U011
Record Dates: First submitted 2023-06-13; First posted 2023-06-23 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-01

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- open-label (Other): UNEEG EpiSight solution
  Interventions: Device: UNEEG EpiSight solution

INTERVENTIONS:
Device: UNEEG EpiSight solution — Implantation subcutis under local anesthetics

SUMMARY:
The present study is a 13 months pre-market open-label, prospective study for confirmation of continuous performance and safety of UNEEG EpiSight solution in subjects with uncontrolled epilepsy (indicated for EEG monitoring with the Implant) in which seizures are detectable in an area of the Implant. The surgical procedure, device satisfaction, and effectiveness of the UNEEG EpiSight solution will also be evaluated during the clinical investigation.

DETAILED DESCRIPTION:
The study is a multi-center study with 2-5 European sites in 2-4 countries. Each site will enrol up to 10 subjects, but total enrolment will not exceed 22 to reach 19 completers of 40 days of recording. The total recruitment period is expected to be 6 months and the total study duration is expected to be approximate 22 months (first subject first visit to last subject out).

ELIGIBILITY:
Inclusion Criteria:

* Patients with uncontrolled epilepsy in which seizures are detectable in an area covered by the implant
* Adults (above 18 years)
* Is willing and able to use the UNEEG EpiSight solution day and night for the duration of the study
* Subject is willing and able to provide written informed consent
* Subject is able to complete all study-required procedures, assessments and follow-up

Exclusion Criteria:

* Vulnerable subjects, including severe cognitive impairment precluding informed consent
* Cannot or do not have the necessary assistance, to properly operate the system
* High risk of surgical complications, such as active systemic infection and haemorrhagic disease
* Involved in therapies with medical devices that deliver electrical energy into the area around the implant, such as cochlear implant(s), implantable brain stimulation and external/transcranial brain stimulation
* Contraindications to the local anaesthetic used during implantation and explantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Usage of UNEEG EpiSight Recorder | Throughout the run of the investigation (enrollment per subject is up to 12 months)
  Number of recording hours by UNEEG EpiSight Recorder per day (24 hours) after 40 days recording

SECONDARY OUTCOMES:
Device deficiencies | Throughout the run of the investigation (enrollment per subject is up to 12 months)
  Nature and frequency of device deficiencies
Adverse events | Throughout the run of the investigation (enrollment per subject is up to 12 months)
  Nature and frequency of adverse events

OTHER OUTCOMES:
Performance | Throughout the run of the investigation (enrollment per subject is up to 12 months)
  Number of recording hours by UNEEG EpiSight solution per day (24 hours) throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Norman Delanty, Prof, Principal Investigator — Beaumont Hospital, Dublin; Daniel Costello, Prof, Principal Investigator — Cork University Hospital; Christoph Beier, Prof, Principal Investigator — Odense University Hospital; Lis Gregoretti Pluss, M.D., Principal Investigator — Regional Hospital of Viborg; Kimmo Jensen, Prof, Principal Investigator — Aalborg University Hospital
Locations (5):
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Odense University Hospital, Odense
  - Regional Hospital of Viborg, Viborg
- Ireland (2):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin

IPD SHARING:
Plan to Share IPD: No